CLINICAL TRIAL: NCT02693704
Title: Evaluation of a Binaural Spatialization Method for Hearing Aids, in Terms of Speech Intelligibility, Speaker Localization and Subjective Preference.
Brief Title: Evaluation of a Binaural Spatialization Method for Hearing Aids
Acronym: BHA(L&S)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Principal Investigator, Gilles Courtois, PhD Student, Sonova AG
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BHALS - 001
Record Dates: First submitted 2016-02-17; First posted 2016-02-29 (Estimated); Results first posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal hearing (Experimental): People showing no hearing loss (< 20 dB HL). Introduction of speech signal via the DAI of two hearing aids Phonak Naida IX SP.
  Interventions: Device: Hearing Aids
- Moderate hearing impaired (Experimental): Patients showing moderate hearing loss (40-60 dB HL).
  Introduction of speech signal via the DAI of two hearing aids among:
  PhonakAudéo V-13 Phonak Baseo Q-P, Q-SP, Q-M13 Phonak Bolero Q-P, Q-SP, Q-M13, Boléro V-P, V-SP Phonak Naida Q-CRT, Q-SP, Q-UP Phonak Sky Q-RIC, Q-SP, Q-UP, Q-M13 Phonak Ambra microP, SP, M H20 Phonak Cassia microP, SP, M H20 Phonak Dalia microP, SP, M H20 Phonak Naida S SP, S UP, S CRT Phonak Solana microP, SP, M H20 Phonak Certéna micro, Art M, Art P, Art SP, Art micro Phonak Exélia micro, Art M, Art P, Art SP, Art micro Phonak Milo Plus micro, Plus SP, Plus UP Phonak Naida SP, SP Junior, UP, UP Junior Phonak Nios micro, S H20 Phonak Versata micro, Art M, Art P, Art SP, Art micro
  Interventions: Device: Hearing Aids
- Severe hearing impaired (Experimental): Patients showing severe hearing loss (60-80 dB HL).
  Introduction of speech signal via the DAI of two hearing aids among:
  PhonakAudéo V-13 Phonak Baseo Q-P, Q-SP, Q-M13 Phonak Bolero Q-P, Q-SP, Q-M13, Boléro V-P, V-SP Phonak Naida Q-CRT, Q-SP, Q-UP Phonak Sky Q-RIC, Q-SP, Q-UP, Q-M13 Phonak Ambra microP, SP, M H20 Phonak Cassia microP, SP, M H20 Phonak Dalia microP, SP, M H20 Phonak Naida S SP, S UP, S CRT Phonak Solana microP, SP, M H20 Phonak Certéna micro, Art M, Art P, Art SP, Art micro Phonak Exélia micro, Art M, Art P, Art SP, Art micro Phonak Milo Plus micro, Plus SP, Plus UP Phonak Naida SP, SP Junior, UP, UP Junior Phonak Nios micro, S H20 Phonak Versata micro, Art M, Art P, Art SP, Art micro
  Interventions: Device: Hearing Aids
- Profound hearing impaired (Experimental): Patients showing profound hearing loss (> 80 dB HL).
  Introduction of speech signal via the DAI of two hearing aids among:
  PhonakAudéo V-13 Phonak Baseo Q-P, Q-SP, Q-M13 Phonak Bolero Q-P, Q-SP, Q-M13, Boléro V-P, V-SP Phonak Naida Q-CRT, Q-SP, Q-UP Phonak Sky Q-RIC, Q-SP, Q-UP, Q-M13 Phonak Ambra microP, SP, M H20 Phonak Cassia microP, SP, M H20 Phonak Dalia microP, SP, M H20 Phonak Naida S SP, S UP, S CRT Phonak Solana microP, SP, M H20 Phonak Certéna micro, Art M, Art P, Art SP, Art micro Phonak Exélia micro, Art M, Art P, Art SP, Art micro Phonak Milo Plus micro, Plus SP, Plus UP Phonak Naida SP, SP Junior, UP, UP Junior Phonak Nios micro, S H20 Phonak Versata micro, Art M, Art P, Art SP, Art micro
  Interventions: Device: Hearing Aids

INTERVENTIONS:
Device: Hearing Aids — The only intervention consists in applying a specific processing on some recorded speech signals, and comparing the performance obtained with such processed samples with ones that have not been processed. The applied processing is a binaural spatialization method that consists in filtering an original audio signal to get a left and right versions (for the two ears). The binaural rendering gives the impression that the speech signal (and thus the speaker) is located in a desired position in the environment.
  Other Names: Hearing instruments

SUMMARY:
This study investigates the possible benefits of using binaural spatialization techniques in digital wireless microphone systems for hearing aids. Speech intelligibility tests, speaker localization tests and preference tests are performed. The results of a diotic (current rendering) and a binaural (suggested rendering) rendering are compared.

DETAILED DESCRIPTION:
The signal processing laboratory (LTS2) of the Swiss Federal Institute of Technology (EPFL) has developed a new feature of sound rendering in hearing aids. This is a collaboration between EPFL and the Swiss company Phonak Communications AG. The new functionality works with the range of Roger products from Phonak, a new generation of FM systems that use a digital transmission.

FM technology refers to a type of wireless system that helps people better understand speech in noisy situations. FM systems commonly work together with a user's hearing aids, although systems are also available for those with otherwise normal hearing (such as people who suffer from APD, ADHD etc.). An FM system works like this: the person speaking wears or holds a transmitter microphone, or the transmitter is placed in the middle of the group (picking up speech from all around). Using harmless radio waves, the FM system sends speech signal(s) to the listener, who wears a tiny FM receiver behind the ear.

The new feature of such systems performs processing of the speaker's speech signal so that it renders information related to their spatial location. This so-called sound "spatialization" is a natural property of the human binaural auditory system, which allows us to localize sounds. However, this sound spatialization is not delivered by the current FM systems. Thanks to the new technology from EPFL and Phonak, it is now possible to include a binaural spatialization of the speech signal in the Roger product of Phonak hearing devices.

ELIGIBILITY:
Inclusion Criteria

* French-native speakers and adults.
* Normal otoscopy.
* No conductive pathology.
* Normal hearing, or moderate to severe, sloping or flat, symmetrical hearing loss.
* User of bilateral Phonak hearing aids, for more than 6 months (hearing-impaired only).

Exclusion Criteria:

* History of tinnitus or hyperacusis.
* Visual impairment, after correction with glasses or not.
* History of chronic or terminal illness or psychiatric disturbance,.
* History of epilepsy or other reactions associated with the proximity to a video screen.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Courtois, Enginner, Principal Investigator — Sonova AG
Locations (1):
- Ecole Polytechnique Fédérale de Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Courtois G, Lissek H, Estoppey P, Oesch Y, Gigandet X. Effects of Binaural Spatialization in Wireless Microphone Systems for Hearing Aids on Normal-Hearing and Hearing-Impaired Listeners. Trends Hear. 2018 Jan-Dec;22:2331216517753548. doi: 10.1177/2331216517753548. PMID 29457537

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Hearing | Moderate Hearing Impaired | Severe Hearing Impaired | Profound Hearing Impaired
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hearing | Moderate Hearing Impaired | Severe Hearing Impaired | Profound Hearing Impaired | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 4 | 9 | 29
  >=65 years | 0 | 4 | 6 | 1 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (2) | 51 (24) | 63 (20) | 38 (18) | 43 (23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 5 | 6 | 19
  Male | 5 | 7 | 5 | 4 | 21
Region of Enrollment [Number; unit: participants]
  Switzerland | 10 | 10 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Speech Intelligibility
Description: Speech recognition score (%) For each group: average of the SRS over all subjects in the group. The SRS correspond to the number of understood words in a sequence of sentences (French HINT database) mixed with several level of masking noise (speech-shaped noise). Some are played diotically, the other are spatialized in various directions. The goal is to ensure that the spatialization processing does not degrade the understanding of the speech.
Time Frame: 1 day of the experiment
Measure: Mean (Standard Deviation); unit: Percentage of understood word
Arm/Group | Normal Hearing | Moderate Hearing Impaired | Severe Hearing Impaired | Profound Hearing Impaired
Number analyzed (Participants) | 10 | 10 | 10 | 10
Percentage of understood word
  Diotic Rendering | 63 (4) | 60 (6) | 59 (6) | 48 (12)
  Spatialized rendering | 68 (3) | 67 (6) | 66 (7) | 47 (9)

2. Primary Outcome: Speaker's Localization
Description: Localization error (in number of spatial sectors)
  For each group: average localization error over all subjects in the group. It is the difference between the actual spatial sector and the one reported by the listeners. There were 5 spatial sectors, and 9 possible locations. For instance: if the stimuli is played in sector 4, and the listener perceives it in 2, then the localization error is |4-2| = 2. The goal is to compare the localization error in 3 conditions: 1/ with no hearing aids (reference of natural localization) and no spatialization 2/ with hearing aids and standard fittings and no spatialization, and 3/ with spatialization applied.
Time Frame: 1 day of the experiment
Measure: Mean (Standard Deviation); unit: Localization error (# spatial sectors)
Arm/Group | Normal Hearing | Moderate Hearing Impaired | Severe Hearing Impaired | Profound Hearing Impaired
Number analyzed (Participants) | 10 | 10 | 10 | 10
Localization error (# spatial sectors)
  Unaided localization | 0.13 (0.04) | 0.45 (0.11) | 0.5 (0.06) | 2.02 (0.38)
  Aided localization | 0.3 (0.1) | 0.33 (0.08) | 0.57 (0.07) | 1.74 (0.34)
  Spatialized localization | 0.45 (0.09) | 0.54 (0.08) | 0.75 (0.21) | 1.65 (0.40)

3. Primary Outcome: Listener's Subjective Preference
Description: Listeners compare two audiovisual stimuli (diotic and spatialized) and Indicate their preference between binaural diotic (no spatialization), spatialized stimuli, or no preference. Results are given as the percentage of participant for the 3 possible answers in each group.
Time Frame: 1 day of the experiment
Measure: Number; unit: Percentage of participants
Arm/Group | Normal Hearing | Moderate Hearing Impaired | Severe Hearing Impaired | Profound Hearing Impaired
Number analyzed (Participants) | 10 | 10 | 10 | 10
Percentage of participants
  Diotic | 60 | 50 | 45 | 30
  Spatialization | 35 | 35 | 40 | 50
  No preference | 5 | 15 | 15 | 20

ADVERSE EVENTS:
Arm/Group | Normal Hearing | Moderate Hearing Impaired | Severe Hearing Impaired | Profound Hearing Impaired
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No